CLINICAL TRIAL: NCT05064371
Title: Interventional, Open-label, Fixed-dose, Long-term Extension Study to Evaluate Safety of Eptinezumab as Preventive Treatment in Patients With Migraine
Brief Title: Long-Term Extension Study With Eptinezumab as Preventive Treatment in Participants With Migraine in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19140B
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — eptinezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eptinezumab (Experimental): Participants will receive eptinezumab 100 milligrams (mg) at the Baseline visit (Week 0) and eptinezumab 100 mg or 300 mg (depending upon the treatment response) at Weeks 12, 24, 36, and 48 by intravenous (IV) infusions.
  Interventions: Drug: Eptinezumab

INTERVENTIONS:
Drug: Eptinezumab — Concentrate for solution for IV infusion

SUMMARY:
This study is an open label extension study, which means that the participants from the Lead-in Study 19140A (NCT04921384) can join this study, if they meet the study Eligibility Criteria, and continue to receive the study drug eptinezumab. The main goal of this study is to investigate long-term safety and tolerability of eptinezumab in Japanese migraine participants.

DETAILED DESCRIPTION:
The total study duration from the Baseline Visit to the Safety Follow-up Visit is approximately 68 weeks and includes an Open-Label Treatment Period (60 weeks) and a Safety Follow-up Period (8 weeks).

ELIGIBILITY:
Key Inclusion Criteria:

* The participant has completed the Primary Outcome Visit (Visit 5) of the lead-in Study 19140A immediately prior to enrolment into this study.
* The participant is indicated for 60-week preventive treatment of chronic migraine with eptinezumab according to the clinical opinion of the investigator.

Key Exclusion Criteria:

* The participant has a serious adverse event (SAE) or a moderate or severe ongoing AE from the Lead-In study considered a potential safety risk by the investigator.
* The participant has a clinically relevant change in vital signs or electrocardiogram (ECG) from the Lead-In study considered a potential safety risk by the investigator.
* The participant has a disease or takes medication that could, in the investigator's opinion, interfere with the assessments of safety, tolerability, or efficacy, or interfere with the conduct or interpretation of the study.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2024-06-08 (Actual); Study Completion 2024-06-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | From Baseline to Week 68

SECONDARY OUTCOMES:
Change From Baseline in the Number of Monthly Migraine Days | Baseline, Week 60
Response: Number of Participants With ≥50% Reduction From Baseline in Monthly Migraine Days (MMDs) | Baseline to Week 60
Change From Baseline in the Headache Impact Test (HIT-6) Score | Baseline, Week 60
Change From Baseline in the Health-Related Quality of Life (EQ-5D-5L) Visual Analogue Scale (VAS) Score | Baseline, Week 60
Patient Global Impression of Change (PGIC) Score | Baseline to Week 60
Change From Baseline in the Most Bothersome Symptom (MBS) Score | Baseline, Week 60

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (17):
- Japan (17):
  - DOI Clinic Internal Medicine, Hiroshima-Shi Naka-Ku, Hiroshima
  - Jinnouchi Neurosurgery Clinic, Kasuga-Shi, Hukuoka
  - Ikeda Neurosurgical Clinic, Kasuga-Shi, Hukuoka
  - Mito Kyodo General Hospital, Mito, Ibaraki
  - Iwate Medical University Uchimaru Medical Center, Morioka, Iwate
  - Atsuchi Neurosurgery Hospital, Kagoshima, Kagoshima-ken
  - Shin Matsudakai Atago Hospital, Kochi, Kôti
  - Sendai Headache and Cranial Nerves Clinic, Sendai-Shi Taihaku-Ku, Miyagi
  - Saitama Neuropsychiatric Institute, Saitama-Shi, Saitama
  - Moriyama Neurological Center Hospital, Edogawa-Ku, Tokyo
  - Tokyo headache clinic, Shibuya-Ku, Tokyo
  - Nagamitsu Clinic, Hofu-Shi, Yamaguchi
  - Tatsuoka Neurology Clinic, Kyoto Shimojo-ku
  - Dokkyo Medical University Hospital, Mibu-machi
  - Japanese Red Cross Shizuoka Hospital, Shizuoka
  - Toyota Memorial Hospital, Toyota-shi
  - Tominaga Hospital, Osaka, Ã"saka